CLINICAL TRIAL: NCT06289855
Title: Impulse Control Disorder Among Parkinson's Disease Patients; Clinical and Neurophysiological Study
Brief Title: Impulse Control Disorder Among Parkinson's Disease Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Roaa Almoataz Abdelrazik Zohni Elsabrout, Assisstant lecturer, neurology department, Assiut university, Assiut University
Other Study IDs: Parkinson's disease
Record Dates: First submitted 2024-02-26; First posted 2024-03-04 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: MDS-UPDRS — Movement disorder society- unified Parkinson disease rating scale (MDS-UPDRS) for Parkinson's disease.
  Movement disorder society- non motor rating scale (MDS-NMS) Cognitive assessment using Scales for Outcomes in Parkinson's disease-Cognition (SCOPA-Cog)
  Using Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale:
  Timed up and go: originally aimed to clinically evaluate dynamic balance in elderly people during the performance of a task MR imaging of the brain will be performed with a 1.5T MR imaging scanner Assessment of Cortical excitability and unhibition by NIHON KOHDEN- neuropack2
  Other Names: MDS-NMS; SCOPA-Cog; Questionnaire for Impulsive-Compulsive Disorders in Parkinson's Disease Rating Scale; Timed up and go; MR imaging of the brain; cortical excietability

SUMMARY:
The goal of this observational study is to learn about impulse control disorders in Parkinson's disease patients.

The main question: it aims to answer:

* Detect Relative frequency of impulse control disorder among Parkinson's disease patients
* Detect Relation between impulse control disorders, and other non motor and motor symptoms in Parkinson's disease patients, using clinical, neurophysiological and radiological assessment

DETAILED DESCRIPTION:
Parkinson disease (PD), is a multisystem disease with motor and non-motor (NM) deficits. Dementia and mild forms of cognitive impairment as well as neuropsychiatric symptoms (i.e., impulse control disorders) are frequent and disabling non-motor symptoms of Parkinson's disease (PD). According to the fifth edition of the American Psychiatric Association's Diagnostic and Statistical Manual (DSM-5), impulse control disorders are defined as "disruptive, impulse-control, while conduct disorders include conditions involving problems in the self-control of emotions and behaviors".

Many studies have highlighted potential risk factors for these behaviors, including the fact that that ICDs are associated with younger age, male sex and younger age at disease onset. Also these behaviors have been consistently linked to the use of dopaminergic medications used to treat Parkinson's disease motor symptoms (dopamine agonists, levodopa, and other agents) and less consistently to neuro-modulation techniques such as deep brain stimulation (DBS).

Up to 14-17% of patients with Parkinson's disease display a set of impulsive-compulsive spectrum disorders during the course of illness. Once uncontrolled behaviors develop, either patients fail understand or recognize the severity of their actions or hide them in shame with devastating social and financial results for themselves and their families.

Previous neuropsychological studies have also demonstrated that impulse control disorders in Parkinson's disease are associated with an altered cognitive profile, characterized by impaired cognitive flexibility and planning capability as well as by more inappropriate behavior and poor feedback processes. Also, Cognitive impairment and dementia in particular are associated with adverse outcomes, including gait impairment and falls, greater disability and caregiver burden, higher economic costs, and increased mortality.

Motor deficits have been repeatedly associated with changes in the activity of the motor cortex, in patients with Parkinson's disease. A key regulator of cortical motor output is the balance between excitation and inhibition, which can be assessed in humans with transcranial magnetic stimulation (TMS) techniques.

A common measure to explore inhibitory mechanisms is the short-interval intracortical inhibition (SICI) induced by paired-pulse TMS stimuli. Several studies have described reduced SICI (i.e. less inhibition) in the motor cortex of patients with Parkinson's disease.

The development of neuroimaging techniques, including Voxel-based morphometry (VBM), which is an automated quantitative magnetic resonance imaging (MRI) technique extensively used to assess the grey matter (GM) morphology changes in the brain and has been widely used in Parkinson's disease. The majority of the studies focused on grey matter (GM) changes in Parkinson's disease associated with motor and non-motor symptoms.

Reduced cortical thickness of fronto-striatal regions has been reported as the key feature to differentiate Parkinson's disease with impulse control disorders from Parkinson's disease without impulse control disorders patients, but a concomitant increased amygdala volume and a positive relationship between impulse control disorders severity and middle frontal and parietal cortical volumes have been also shown. In addition, two studies showed an increased cortical thickness in meso-limbic regions and another one reported a relatively preserved grey matter in Parkinson's disease with impulse control disorders patients compared with Parkinson's disease without impulse control disorders cases. Also studies showed that changes in grey matter volume are associated with lack of inhibition related to impulse control disorders behaviors in Parkinson's disease.

Therefore; impulse control disorder is becoming an increasingly recognized psychiatric complication in Parkinson's disease; and whether or not it's associated with cortical dysfunction, and further cognitive and gait and balance affection, need further clinical, neurophysiological and radiological analysis, to further understand the underlying mechanism.

ELIGIBILITY:
1. Inclusion criteria:

   * The study will include patients with Parkinson's disease, diagnosed according to the UK Parkinson's Disease Society Brain Bank criteria. (16)
   * Bradykinesia (slowness of initiation of voluntary movements with progressive reduction in speed and amplitude of repetitive actions).
   * And at least one of the following: Muscular rigidity, 4-6 Hz rest tremor Postural instability not caused by primary visual, vestibular, cerebellar or proprioceptive dysfunction
2. Exclusion criteria:

   * History of strokes with stepwise progression of Parkinsonian features.
   * History of head injury.
   * History of definite encephalitis.
   * Oculogyric crises.
   * Neuroleptic treatment at onset of symptoms.
   * Strictly unilateral features after three years.
   * Supranuclear gaze palsy.
   * Cerebellar signs.
   * Early severe autonomic involvement.
   * Early severe dementia with disturbances of memory, language and praxis.
   * Babinski sign.
   * Presence of a cerebral tumor or communicating hydrocephalus on CT scan.
   * Negative response to large doses of levodopa (if malabsorption excluded).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Parkinson's disease attending Assiut University neurology outpatient clinic and internal department
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-08-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
number of patients with impulse control disorder among Parkinson's disease patients | 1 year
  Relative frequency of impulse control disorder among Parkinson's disease patients, and comparing those with impulse control and those without impulse control disorder, clinically and neurophysiologically

SECONDARY OUTCOMES:
percent of cognition affection, gait affection among patients with impulse control disorder among Parkinson's disease patients | 1 year
  Relation between impulse control disorders, other non motor and motor symptoms in Parkinson's disease patients, using clinical, neurophysiological and radiological assessment
volume of cortex and basal ganglia in patients with impulse control disorder among Parkinson's disease patients | 1 year
  detect cortical and subcortical volume by MRI volumetry
cortical excitability and inhibition inpatients with impulse control disorder among Parkinson's disease patients | 1 year
  neurophysiological assessment of cortical excitability

IPD SHARING:
Plan to Share IPD: No
The confidentiality of patient's information will be maintained throughout the study, only clinical data will be shared

REFERENCES:
- [Result] Martin-Bastida A, Delgado-Alvarado M, Navalpotro-Gomez I, Rodriguez-Oroz MC. Imaging Cognitive Impairment and Impulse Control Disorders in Parkinson's Disease. Front Neurol. 2021 Nov 5;12:733570. doi: 10.3389/fneur.2021.733570. eCollection 2021. PMID 34803882
- [Result] Jellinger KA. Neuropathobiology of non-motor symptoms in Parkinson disease. J Neural Transm (Vienna). 2015 Oct;122(10):1429-40. doi: 10.1007/s00702-015-1405-5. Epub 2015 May 15. PMID 25976432
- [Result] Weintraub D, Koester J, Potenza MN, Siderowf AD, Stacy M, Voon V, Whetteckey J, Wunderlich GR, Lang AE. Impulse control disorders in Parkinson disease: a cross-sectional study of 3090 patients. Arch Neurol. 2010 May;67(5):589-95. doi: 10.1001/archneurol.2010.65. PMID 20457959
- [Result] Cossu G, Rinaldi R, Colosimo C. The rise and fall of impulse control behavior disorders. Parkinsonism Relat Disord. 2018 Jan;46 Suppl 1:S24-S29. doi: 10.1016/j.parkreldis.2017.07.030. Epub 2017 Aug 1. PMID 28818561
- [Result] Grassi G, Albani G, Terenzi F, Razzolini L, Ramat S. New pharmacological and neuromodulation approaches for impulsive-compulsive behaviors in Parkinson's disease. Neurol Sci. 2021 Jul;42(7):2673-2682. doi: 10.1007/s10072-021-05237-8. Epub 2021 Apr 14. PMID 33852081
- [Result] Probst CC, van Eimeren T. The functional anatomy of impulse control disorders. Curr Neurol Neurosci Rep. 2013 Oct;13(10):386. doi: 10.1007/s11910-013-0386-8. PMID 23963609
- [Result] Menon V. Large-scale brain networks and psychopathology: a unifying triple network model. Trends Cogn Sci. 2011 Oct;15(10):483-506. doi: 10.1016/j.tics.2011.08.003. Epub 2011 Sep 9. PMID 21908230
- [Result] Lichter DG, Benedict RHB, Hershey LA. Importance of Balance-Gait Disorder as a Risk Factor for Cognitive Impairment, Dementia and Related Non-Motor Symptoms in Parkinson's Disease. J Parkinsons Dis. 2018;8(4):539-552. doi: 10.3233/JPD-181375. PMID 30124451
- [Result] Hyland BI, Seeger-Armbruster S, Smither RA, Parr-Brownlie LC. Altered Recruitment of Motor Cortex Neuronal Activity During the Grasping Phase of Skilled Reaching in a Chronic Rat Model of Unilateral Parkinsonism. J Neurosci. 2019 Nov 27;39(48):9660-9672. doi: 10.1523/JNEUROSCI.0720-19.2019. Epub 2019 Oct 22. PMID 31641050
- [Result] Ammann C, Dileone M, Pagge C, Catanzaro V, Mata-Marin D, Hernandez-Fernandez F, Monje MHG, Sanchez-Ferro A, Fernandez-Rodriguez B, Gasca-Salas C, Manez-Miro JU, Martinez-Fernandez R, Vela-Desojo L, Alonso-Frech F, Oliviero A, Obeso JA, Foffani G. Cortical disinhibition in Parkinson's disease. Brain. 2020 Dec 5;143(11):3408-3421. doi: 10.1093/brain/awaa274. PMID 33141146
- [Result] Bologna M, Guerra A, Paparella G, Giordo L, Alunni Fegatelli D, Vestri AR, Rothwell JC, Berardelli A. Neurophysiological correlates of bradykinesia in Parkinson's disease. Brain. 2018 Aug 1;141(8):2432-2444. doi: 10.1093/brain/awy155. PMID 29901693
- [Result] Guerra A, Suppa A, D'Onofrio V, Di Stasio F, Asci F, Fabbrini G, Berardelli A. Abnormal cortical facilitation and L-dopa-induced dyskinesia in Parkinson's disease. Brain Stimul. 2019 Nov-Dec;12(6):1517-1525. doi: 10.1016/j.brs.2019.06.012. Epub 2019 Jun 11. PMID 31217080
- [Result] Casarotto S, Turco F, Comanducci A, Perretti A, Marotta G, Pezzoli G, Rosanova M, Isaias IU. Excitability of the supplementary motor area in Parkinson's disease depends on subcortical damage. Brain Stimul. 2019 Jan-Feb;12(1):152-160. doi: 10.1016/j.brs.2018.10.011. Epub 2018 Oct 23. PMID 30416036
- [Result] Zhai H, Fan W, Xiao Y, Zhu Z, Ding Y, He C, Zhang W, Xu Y, Zhang Y. Voxel-based morphometry of grey matter structures in Parkinson's Disease with wearing-off. Brain Imaging Behav. 2023 Dec;17(6):725-737. doi: 10.1007/s11682-023-00793-3. Epub 2023 Sep 22. PMID 37735325
- [Result] Tessitore A, Santangelo G, De Micco R, Vitale C, Giordano A, Raimo S, Corbo D, Amboni M, Barone P, Tedeschi G. Cortical thickness changes in patients with Parkinson's disease and impulse control disorders. Parkinsonism Relat Disord. 2016 Mar;24:119-25. doi: 10.1016/j.parkreldis.2015.10.013. Epub 2015 Oct 20. PMID 26810913